CLINICAL TRIAL: NCT06281145
Title: A Study on Therapeutic Potential of Stress-Reducing Intervention in Patients With Solid Tumors
Brief Title: Stress-Reducing Intervention in Patients With Colorectal and Breast Cancer
Acronym: SRI-BrCa_CRC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Comenius University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RSV-SK001/UC-SK004/OUSA
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Colon Cancer
Keywords: Colon Cancer; Invasive Breast Cancer; Neoadjuvant Chemotherapy; Standard of Care; Inflammation; Stress; Telemedicine; Circadian rhythms; Sleep Quality; Quality of Life; Autonomic Nervous System; Heart-Rate Variability
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Inflammation; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The study consists of two cohorts (breasts cancer and colorectal cancer) with two arms SOC + intervention vs SOC alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care + HRV biofeedback intervention (Experimental): Experimental: Heart-rate variability (HRV) biofeedback intervention + standard of care Deep paced breathing with the HRV monitoring performed three times a day for seven minutes during three months with standard of care.
  Cohort A- breast cancer, Cohort B- colon cancer
  Interventions: Behavioral: Heart-rate variability biofeedback intervention
- Standard of care (No Intervention): Cohort A- neoadjuvant chemotherapy +/- targeted therapy +/- immunotherapy defined standard of care in current European Society For Medical Oncology (ESMO) guideline in the defined disease subtype Cohort B- adjuvant chemotherapy +/- targeted therapy +/- immunotherapy defined standard of care in current ESMO guideline in the defined disease subtype

INTERVENTIONS:
Behavioral: Heart-rate variability biofeedback intervention — Daily deep paced breathing 3-times (minimum 7 minutes each) for 3 months
  Arms: Standard of care + HRV biofeedback intervention

SUMMARY:
The goal of this interventional study is to test the heart-rate variability biofeedback intervention (HRV BI) in 2 cohorts of patients. Cohort A will evaluate the effect of the addition of HRV BI in patients with breast cancer treated in the neoadjuvant setting (vs. standard of care alone, SOC) followed by local therapy (surgery +/-radiotherapy). Cohort B will evaluate the effect of the addition of HRV BI in patients with colon cancer after surgery in the adjuvant setting (vs. standard of care alone, SOC).

DETAILED DESCRIPTION:
This is a prospective, interventional, clinical study with in 2 cohorts. Target of subjects is 50 per cohort and an anticipated total duration of 36 months.

Participants will undergo 4 sessions of HRV BI with the trainer where they will learn about the prognostic role of the vagal nerve in cancer and in reducing distress and pain, and how to perform deep paced breathing with the HRV monitoring. They will perform the training daily (3-times, minimum 7 minutes each) at home with the online control for 3 months.

Researchers will compare the effect of addition of 3-months training of HRV BI to SOC on inflammation, HRV, quality of life (QoL), cognitive functions, salivary cortisol slopes, sleep quality and treatment outcomes of patients with colorectal and breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years.
2. Pathologically confirmed breast cancer indicated for neoadjuvant systemic treatment or colon cancer after curative surgery indicated for adjuvant systemic treatment.
3. Adequate renal functions: measured or calculated (by Cockcroft formula) creatinine clearance > 60 ml/min.
4. Absolute granulocytes count ≥ 1,500/mm3, platelets ≥ 100,000 mm3, bilirubin ≤ 1.5x the upper limit of normal value.
5. Adequate liver functions defined by AST (Aspartate aminotransferase) and ALT (Alanine transaminase) ≤ 3xUNL (upper normal of limit).
6. Basic computer skills of patient or his family member.
7. Signed informed consent.

Exclusion Criteria:

1. Previous chemotherapy.
2. Previous malignancy, except for basal-cell carcinoma of the skin within last 5 years.
3. Patients with know primary immunodeficiency and patients infected by the Human Immunodeficiency Virus (HIV).
4. Patient receiving long term corticosteroid treatment, anti-arrhythmic drugs and opioids who can not withdraw the treatment for the period of application of the heart rate variability (HRV) biofeedback training.
5. Patients with diabetes mellitus, cardiac arrhythmia, cardiac pacemaker implant.
6. Patients who do not fit inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2029-03-15 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint - inflammation | 36 months
  he effect of 3-month heart rate variability (HRV) biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on inflammation (IL-6, Tumor necrosis factor α, IL-10 from peripheral blood sample in pg/ml and tumour infiltrating lymphocytes (TIL) in %).
Primary endpoint - QoL | 36 months
  Effect of HRV biofeedback training on quality of life (HRV biofeedback + SOC, vs. The effect of 3-month heart rate variability (HRV) biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on EORTC-QLQ-C30 (version 3) score (QLQ- Quality Life Questionnaire). The EORTC-QLQ-C30 has 30 items divided into five functional scales (physical, role, cognitive, emotional, and social), and three symptom scales (fatigue, pain, and nausea and vomiting). The score for each scale as well as the sum score for the whole instrument is standardized to values 0 to 100, with a higher score meaning a worse outcome.
Primary endpoint - executive functions | 36 months
  Effect of HRV biofeedback training on executive functions (HRV biofeedback + SOC, vs. SOC alone) measured by Stroop task mean response time for color-word condition.
Primary endpoint- salivary cortisol slopes | 36 months
  The effect of 3-month heart rate variability (HRV) biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on salivary cortisol slopes (difference between bedtime and awakening saliva cortisol concentration in ng/ml).
Primary endpoint- sleep quality | 36 months
  The effect of 3-month heart rate variability (HRV) biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on sleep quality measured by both actigraphy and self-report data. The main variables are total time spent sleeping (in hours and minutes), and sleep efficiency (proportion of time spent sleeping vs. time spent in bed trying to sleep).
Primary endpoint - heart rate variability (HRV) | 36 months
  Effect of HRV biofeedback training on HRV indexed by the root mean square of successive differences between heartbeats (RMSSD) in ms.
Primary endpoint - Working memory | 36 months
  The effect of 3-month heart rate variability (HRV) biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on working memory measured by digit span test score (the number of remembered digits in the longest passed sequence), for both forward and backward condition.

SECONDARY OUTCOMES:
Secondary endpoint - Pathologic Complete Response (pCR) and Residual Cancer Burden (RCB) rate in cohort A | 36 months
  The effect of 3-month heart rate variability (HRV)biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on pCR rate evaluated pathologically in surgical specimen after neoadjuvant therapy, value pCR, RCB I, RCB II, RCB III.
Secondary endpoint - Relapse-free Survival (RFS) | 60 months
  The effect of 3-month heart rate variability (HRV) biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on RFS for cohort A and B measured in months from the day of curative surgery.
Secondary endpoint - Overall survival (OS) | 96 months
  The effect of 3-month heart rate variability (HRV) biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on OS for cohort A and B measured in months from the day of curative surgery.
Secondary endpoint - Serious Adverse Events (SAE) | 36 months
  The effect of 3-months heart rate variability (HRV) biofeedback training and conventional cancer treatment (standard of care, SOC) vs. SOC alone on serious adverse events (SAEs) of chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Elizabeth Cancer Institute, Bratislava, Slovakia